CLINICAL TRIAL: NCT01032993
Title: Clinical Trial of CoQ10 for Mild-to-Moderate Statin-Associated Muscle Symptoms
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Catherine Buettner (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor-Investigator, Catherine Buettner, Physician, Beth Israel Deaconess Medical Center
Organization: Beth Israel Deaconess Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: K23AR055664 (NIH); K23AR055664 (NIH)
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Results first posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2016-11

CONDITIONS: Pain; Weakness; Cramps; Myalgia or Myositis Nos; HMG COA Reductase Inhibitor Adverse Reaction
Keywords: CoQ10; Statins; Myalgia; Muscle Pain; Muscle Weakness
MeSH Terms: conditions — Pain; Asthenia; Muscle Cramp; Myalgia; Myositis, Inclusion Body; Muscle Weakness | interventions — coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coenzyme Q10 (Active Comparator): 600 mg of CoQ10 taken as 300 mg (three 100 mg wafers) two times daily. Study wafers: ChewQ (Tishcon Corp, Westbury, NY) are chewable wafers each containing 100 mg of Coenzyme Q10 (ubidecarenone USP). All participants randomized continued use of simvastatin 20 mg started during the run-in phase of the study.
  Interventions: Dietary Supplement: Coenzyme Q10
- Placebo (Placebo Comparator): Placebo was manufactured by the manufacturer of ChewQ, Tishcon Corp (Westbury, NY), included the same excipients, but no active CoQ10, and looked and tasted identical to active agent. All participants randomized continued use of simvastatin 20 mg started during the run-in phase of the study.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Coenzyme Q10 — 300 mg of CoQ10 (three 100 mg chewable tablets) 2 times daily for 4 weeks
  Arms: Coenzyme Q10
Other: Placebo — Placebo (three chewable tablets) 2 times daily for 4 weeks
  Arms: Placebo

SUMMARY:
This study will evaluate whether a dietary supplement, coenzyme Q10 (CoQ10), will improve muscle symptoms, such as muscle aches, pains, cramps, and/or weakness, which are experienced by some individuals who use statin medications.

DETAILED DESCRIPTION:
This study will recruit individuals who have had muscle symptoms while using a statin. During the first part of the study, volunteers will be given a statin medication to see if their muscle symptoms return. Those who experience muscle symptoms on this statin rechallenge will be invited to continue in the second part of the trial, in which participants will be randomly assigned to receive either CoQ10 or a placebo (sugar pill) to take with statin medication. We hypothesize that those who receive CoQ10 will experience an improvement in their muscle symptoms compared to those who receive placebo, and, secondarily, that those who receive CoQ10 will be more likely to continue taking the statin medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of muscle symptoms (such as aches, pains, cramps and/or weakness) while taking a statin drug that persisted for at least 2 weeks on a statin

Exclusion Criteria:

* Plasma creatine kinase levels > 3 times the upper normal limit
* Liver enzymes, alanine transferase (ALT) or aspartate transferase (AST) > 2 times the upper normal limit
* Pregnancy or breastfeeding (a contraindication for statin use)
* Severe renal impairment, defined as glomerular filtration rate (GFR) < 30 ml/min/1.73 m2
* Bleeding disorder, current use of warfarin, an international normalized ratio (INR) greater than 1.5, or a platelet count less than 100,000 mm3
* Contraindication to strength testing, including myocardial infarction, unstable angina, or revascularization procedure within the past six weeks, a history of brain aneurysm or stroke
* Chest or abdominal surgery within the past six weeks
* Severe persistent pain related to other causes
* Unable to complete self-administered questionnaires, or unable to read or converse in English

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2009-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Buettner, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No consent for sharing IPD from trial participants was obtained when this clinical trial began

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Persons with a history of statin myalgia were recruited from the greater Boston area using flyers, ads, and announcements to seek volunteers. A history of statin myalgia was defined as having muscle symptoms thought to be due to a statin, with symptoms that began after a statin was started and that persisted for at least 2 weeks while using statin.
Pre-assignment Details: Confirmation of statin myalgia was based on completing a statin washout, and statin rechallenge. On washout, improvement of symptoms within 2 months was required to advance. On rechallenge, simvastatin 20 mg daily was given, and only those with return of symptoms within 3 months were randomized. Out of 68 participants enrolled, 39 were randomized.
Groups:
- Coenzyme Q10: The Coenzyme Q10 arm used 600 mg of CoQ10 taken as 300 mg (three 100 mg wafers) two times daily for 4 weeks. Active study wafers were ChewQ (ubidecarenone) and were manufactured by Tishcon Corp, (Westbury, NY). All participants randomized to either arm were instructed to continue use of simvastatin 20 mg daily
- Placebo: The Placebo arm used placebo wafers taken as three wafers two times daily for 4 weeks. Placebo wafers contained the same excipients as the active wafers, but contained no active CoQ10. The wafers looked and tasted identical to active agent, and were manufactured by the same manufacturer of the active agent, Tishcon Corp (Westbury, NY). All participants randomized to either arm were instructed to continue use of simvastatin 20 mg daily
Period: Overall Study
Arm/Group | Coenzyme Q10 | Placebo
Started | 19 | 20
Completed | 19 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Coenzyme Q10: CoQ10 300 mg 2 x daily + Simvastatin 20 mg daily
- Placebo: Placebo 2 x daily + Simvastatin 20 mg daily
- Total: Total of all reporting groups
Arm/Group | Coenzyme Q10 | Placebo | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (7.9) | 60.1 (11.2) | 61.0 (9.7)
Gender [Count of Participants; unit: Participants]
  Female | 14 | 6 | 20
  Male | 5 | 14 | 19
Race/Ethnicity, Customized [Number; unit: participants]
  Non-Hispanic White | 17 | 17 | 34
  Other | 2 | 3 | 5
Alcohol Servings/Day [Number; unit: participants]
  0 to 1 | 8 | 8 | 16
  2 to 4 | 9 | 9 | 18
  5 or more | 2 | 3 | 5
Exercise [Number; unit: participants]
  Moderate/Vigorous | 10 | 8 | 18
  None/Light | 9 | 12 | 21
Diabetes [Number; unit: participants]
  Yes | 5 | 4 | 9
  No | 14 | 16 | 30
Hypertension [Number; unit: participants]
  Yes | 14 | 16 | 30
  No | 5 | 4 | 9
Pain (baseline) visual analog scale (0-10) [Mean (Standard Deviation); unit: units on a scale] — Pain was rated on a scale from 0 to 10, where 0 =n o pain and 10 = pain as bad as you can imagine
  units on a scale | 4.4 (2.2) | 4.9 (1.9) | 4.6 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Reduction in Muscle Pain Associated With Statin Use
Description: Clinically significant pain reduction was defined, a priori, as a reduction > 1.5 points on the Brief Pain Inventory-Severity Scale (BPI-SS), range: 0 to 10
Time Frame: 4 weeks
Measure: Number; unit: % of participants with pain reduction
Arm/Group | Coenzyme Q10 | Placebo
Number analyzed (Participants) | 19 | 20
% of participants with pain reduction | 53 | 65

2. Secondary Outcome: Continuation of Statin
Description: Adherence of statin use was defined a priori as participant using Simvastatin 20 mg /day at the end of 4 weeks and having used >85% of statin doses.
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | Coenzyme Q10 | Placebo
Number analyzed (Participants) | 19 | 20
participants
  Adherent with Statin at 4 wks | 17 | 18
  Not Adherent with Statin at 4 wks | 2 | 2

3. Secondary Outcome: Percentage of Participants With Improvement in Disability Related to Muscle Pain
Description: Disability improvement was based on patient report of improvement they felt was meaningful to them
Time Frame: 4 weeks
Measure: Number; unit: % reporting improved function
Arm/Group | Coenzyme Q10 | Placebo
Number analyzed (Participants) | 19 | 20
% reporting improved function | 36 | 40

4. Secondary Outcome: Percentage of Participants With Adverse Effects
Description: serious adverse effects and possible side effects were tracked through all phases of the study by participant interview and checklist at each visit, up to 4 weeks.
Time Frame: 4 weeks
Population: 3 serious adverse events occurred during the study that were judged unrelated to the study: specifically, 3 participants were hospitalized prior to randomization, 1 for pneumonia; 1 for a back injury; and 1 for a mental health condition. All recovered. There were no SAE during the randomization period. Non serious AEs are listed below.
Measure: Number; unit: % of participants reporting
Arm/Group | Coenzyme Q10 | Placebo
Number analyzed (Participants) | 19 | 20
% of participants reporting
  Nausea/dyspepsia | 21 | 10
  Fatigue | 10 | 10

ADVERSE EVENTS:
Time Frame: Serious adverse effects and possible side effects were tracked through all phases of the study by participant interview and checklist at each visit, up to 4 weeks.
Description: 3 serious adverse events occurred during the study that were judged unrelated to the study agent. Specifically, 3 participants were hospitalized prior to randomization: 1 for pneumonia; 1 for a back injury; and 1 for a mental health condition. All recovered. There were no SAE during the randomization period. Non serious AEs are listed below.
Arm/Group | Coenzyme Q10 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 4/19 | 2/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coenzyme Q10 (N=19) | Placebo (N=20)
Nausea/dyspepsia (Gastrointestinal disorders) | 4 (4) | 2 (2)
Fatigue (General disorders) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
100 participants were planned to achieve >50 randomized. However, due to slow recruiting, the CoQ10 and placebo expired and we were unable to obtain more. Therefore only 68 participants were enrolled and ultimately 39 participants were randomized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No